CLINICAL TRIAL: NCT06101706
Title: Assessment of Fatigue in Psoriatic Arthritis and Cutaneous Psoriasis Patients
Acronym: RPso-Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RPso-Fatigue
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis; Psoriasis
Keywords: Fatigue; Quality of life
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoriatic arthritis patients (Other)
  Interventions: Behavioral: Fatigue assessment; Behavioral: Quality of life assessment; Other: Assess severity of psoriatic arthritis
- Cutaneous psoriasis patients (Other)
  Interventions: Behavioral: Fatigue assessment; Behavioral: Quality of life assessment; Other: Assess severity of cutaneous psoriasis

INTERVENTIONS:
Behavioral: Fatigue assessment — FACIT-F questionnaire and Visual Analog Scale for fatigue
Behavioral: Quality of life assessment — PsAID-12 questionnaire, DLQI questionnaire and SF-36 questionnaire
Other: Assess severity of psoriatic arthritis — DAPSA score
  Arms: Psoriatic arthritis patients
Other: Assess severity of cutaneous psoriasis — PASI score
  Arms: Cutaneous psoriasis patients

SUMMARY:
Psoriatic arthritis is characterized with pain, swelling and joint stiffness. These are inflammatory reactions against tendons, ligaments and joints associated with fatigue. In France, almost 93.000 people are affected by psoriatic arthritis and the main symptoms appear between 30 and 50 years old. Psoriatic arthritis may be due to a genetic predisposition involving the HLA B27 gene, or to environmental factors such as stress, physical or psychological trauma, or infection. Obesity, type 2 diabetes and hypertension can also be factors associated with the onset of psoriatic arthritis.

Cutaneous psoriasis is a non-contagious chronic inflammatory skin disease, where the skin renews itself at an abnormally rapid rate. In France, between 2 and 3 million people are affected by cutaneous psoriasis, approximately 60.000 new cases every year. The disease begin in adolescence or young adulthood. There are multiples forms of cutaneous psoriasis (plaque, guttate, pustular, erythrodermic, inverse, facial, scalp, nail and mucous membranes). The main symptom is the appearance of thick red patches of varying size, covered with white dead skin. These lesions are most often found on the hands, elbows, knees, lower back, face or scalp. There is little to no itching. During periods of remission, lesions can disappear completely or partially, then reappear during a new attack, called a "flare-up". A familial genetic predisposition is present in 1/3 of psoriasis patients. Other immune and environmental factors, such as medication, irritations, sun exposure or psychological state, can influence psoriasis flare-ups. Psoriasis has no serious health consequences, but it can be aesthetically unpleasant, affect relationships and psychological well-being.

Fatigue is a common symptom in psoriatic arthritis patients, and can significantly affect quality of life and work capacity. Fatigue, which affects over 50% of psoriatic arthritis patients, is a major component of the disease's impact. Fatigue in psoriatic arthritis is a much-discussed topic in the current scientific literature. Although less well documented, patients with cutaneous psoriasis also experience fatigue. Several clinical trials show that, once the disease has been treated, fatigue tends to diminish, but in some cases, the treatment itself may play a role in the vicious fatigue circle. The risk of suffering other skin manifestations despite being under treatment can often be misunderstood by the patient, leading to increased depression and fatigue. Overall, treatments are more likely to play an important role in the variability of fatigue. Ultimately, fatigue is a multifactorial symptom that can be linked either to the disease itself, or to the therapies used. It therefore appears to be the most difficult symptom to treat with commercially available therapies.

As fatigue is a major symptom of psoriatic arthritis and cutaneous psoriasis, it is essential to know how the therapies offered influence this symptom, and to study whether certain therapies are more likely to increase it, despite their efficacy on joint and skin symptoms. It is also relevant to determine whether fatigue is correlated with disease severity, duration and even more so with the therapy used, to better understand the psychological impact of patients with psoriatic arthritis or cutaneous psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient with psoriatic arthritis of any stage or duration, followed in the center's rheumatology or dermatology departments, whether or not treated with systemic therapy.
* Patient with all forms of cuteaneous psoriasis (plaque, inverted, erythrodermic or guttate), whatever the stage or duration of the disease, followed in the center's dermatology department, whether or not treated with systemic therapy.

Exclusion Criteria:

* Patient with auto-inflammatory joint disease: ankylosing spondylitis, rheumatoid arthritis.
* Patient with auto-immune disease involving skin lesions: lupus, dermatomyositis, morphea, pemphigus, pemphigoid, Sjögren's syndrome.
* Cancer.
* Pregnant women.
* Severe heart failure (New York Heart Association Class III or IV).
* Severe renal failure (DFG < 30).
* Hepatic failure.
* Anemia < 10g/dL.
* Patient under legal protection, deprived of liberty or unable to be included in a research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Compare fatigue between psoriatic arthritis and cutaneous psoriasis patients | Baseline
  Functional Assessment of Chronic Illness Therapy System of Quality of Life questionnaire : FACIT-F (this questionnaire contains 13 items, each item score can range from 0 to 5, the total score range from 0 to 52, a high score represents a high quality of life).

SECONDARY OUTCOMES:
Assess and compare fatigue score by disease, treatment type and demographic data | Baseline
  Fatigue will be assessed by Visual Analog Scale (a subjective measure for fatigue, scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no fatigue" and "maximum fatigue imaginable").
Assess and compare quality of life | Baseline
  Psoriatic Arthritis Impact of Disease : PsAID-12 (this questionnaire contains 12 items, the total score range from 0 to 10, a high score represents the worst health condition).
Assess and compare quality of life | Baseline
  Dermatology Life Quality Index : DLQI (this questionnaire contains 10 items, the total score range from 0 to 30, a high score represents a low quality of life).
Assess and compare quality of life | Baseline
  36-Item Short Form Survey : SF-36 (this questionnaire contains 36 items, the total score range from 0 to 100, a high score represents a high quality of life).
Assess severity of psoriatic arthritis | Baseline
  Disease Activity in Psoriatic Arthritis : DAPSA (this score range from 0 to 164, a high score represents a more severe disease).
Assess severity of cutaneous psoriasis | Baseline
  Psoriasis Area Severity Index : PASI (this score range from 0 to 72, a high score represents a more severe disease).

CONTACTS AND LOCATIONS:
Overall Officials: Carina Mihu, Medical Intern, Principal Investigator — Centre Hospitalier d'Avignon, Service de dermatologie
Locations (1):
- Centre Hospitalier d'Avignon, Avignon, France